CLINICAL TRIAL: NCT02370030
Title: Controlled Randomized Multi-centric Clinical Trial on the Effect of Citrulline on the Clinical and Biochemical Evolution of Patients With Sepsis.
Brief Title: Effect of Citrulline on the Clinical and Biochemical Evolution of Patients With Sepsis.
Acronym: CITRUSEP
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, Eduardo Almeida Gutiérrez, Head Researcher, Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R-2014-785-082
Record Dates: First submitted 2015-02-18; First posted 2015-02-24 (Estimated); Last update posted 2015-08-28 (Estimated); Status verified 2015-08

CONDITIONS: Sepsis
Keywords: sepsis; citrulline; endothelial; toxemia; endothelial determination of progression; with vs without citrulline
MeSH Terms: conditions — Sepsis; Toxemia | interventions — citrulline malate; Citrulline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Active Comparator): Oral or nasogastric administration of 10 g citrulline malate daily. Blood and urine samples to determine biomarkers of endothelial damage (IL 6, IL 10 , nitric oxide and microalbuminuria), with a second sampling after 7 days of intervention. Disease severity will be measure with various scales, including APACHE II, SOFA
  Interventions: Dietary Supplement: Citrulline malate
- Placebo (Placebo Comparator): 10 g of maltodextrin will be substituted for the citrulline. Blood and urine samples to determine biomarkers of endothelial damage (IL 6, IL 10 , nitric oxide and microalbuminuria), with a second sampling after 7 days of intervention. Disease severity will be measure with various scales, including APACHE II, SOFA
  Interventions: Dietary Supplement: Citrulline malate

INTERVENTIONS:
Dietary Supplement: Citrulline malate — Active comparator: 10 g/day citrulline malate during 7 days
  Other Names: Citrulline

SUMMARY:
Triple blind placebo-controlled study to determine if administering citrulline in patients with sepsis and severe sepsis slows progression to multiple organ failure and death, measuring biomarkers of endothelial dysfunction. Patients are divided into placebo or citrulline and followed up for 1 month.

DETAILED DESCRIPTION:
Consecutive patients with sepsis are being recited from intensive care unite of IMSS at the CMN Siglo XXI and CMN La Raza over the period of november 2015 through june 2016. After signing an informed consent they will be randomized into 80 for intervention arm and 80 for the placebo arm. All patients will receive usual medical treatment; and during seven days citurlline arm subjects will receive supplementation with oral or nasogastric citrulline (10 g/day), while other group patients will receive during seven days oral or nasogastric placebo (10 g/day) with no visible difference between these. Microalbuminuria and interleukines 1, 6, and 10 will be measured at randomization and at day 7. All subjects will be followed for 28 days, and after the follow-up period results will be analyzed to determine de efficacy and safety of citrulline, primary outcome are the incidence of multiple organic failure and death, also microalbuminuria levels 1,6,10-interleukines. We will use Student-t and Chi2 for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Sepsis
* Severe sepsis
* Diagnosis of sepsis in the first 36 hours of hospitalization.
* Informed Consent
* Intestinal tract intact

Exclusion Criteria:

* Terminal cancer
* Acute and chronic liver diseases
* Chronic renal failure.
* Acute renal failure AKIN III.
* Pregnant and postpartum women
* Dying patients.
* Patients with cardiac arrest.
* Active gastrointestinal bleeding.
* Steroids or immunosuppressants.
* Enrolled in another study intervention.
* Citrulline allergy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2014-11; Primary Completion 2016-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Multiple organ failure | 1 month
  Progression to multiple organ failure ending in death

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Almeida Gutierrez, MSc, Study Director — Coordinación de Investigación en Salud, México.
Locations (2):
- Mexico (2):
  - CME Centro Mèdico Siglo XXI, Mexico City, Mexico City
  - CME La Raza, Mexico City, Mexico City

REFERENCES:
- [Result] Kao CC, Bandi V, Guntupalli KK, Wu M, Castillo L, Jahoor F. Arginine, citrulline and nitric oxide metabolism in sepsis. Clin Sci (Lond). 2009 Jun 2;117(1):23-30. doi: 10.1042/CS20080444. PMID 19105791
- [Result] Barr FE, Tirona RG, Taylor MB, Rice G, Arnold J, Cunningham G, Smith HA, Campbell A, Canter JA, Christian KG, Drinkwater DC, Scholl F, Kavanaugh-McHugh A, Summar ML. Pharmacokinetics and safety of intravenously administered citrulline in children undergoing congenital heart surgery: potential therapy for postoperative pulmonary hypertension. J Thorac Cardiovasc Surg. 2007 Aug;134(2):319-26. doi: 10.1016/j.jtcvs.2007.02.043. PMID 17662768
- [Result] Piton G, Manzon C, Monnet E, Cypriani B, Barbot O, Navellou JC, Carbonnel F, Capellier G. Plasma citrulline kinetics and prognostic value in critically ill patients. Intensive Care Med. 2010 Apr;36(4):702-6. doi: 10.1007/s00134-010-1751-6. PMID 20084502
- [Result] Piton G, Belon F, Cypriani B, Regnard J, Puyraveau M, Manzon C, Navellou JC, Capellier G. Enterocyte damage in critically ill patients is associated with shock condition and 28-day mortality. Crit Care Med. 2013 Sep;41(9):2169-76. doi: 10.1097/CCM.0b013e31828c26b5. PMID 23782971
- [Result] Luiking YC, Poeze M, Ramsay G, Deutz NE. Reduced citrulline production in sepsis is related to diminished de novo arginine and nitric oxide production. Am J Clin Nutr. 2009 Jan;89(1):142-52. doi: 10.3945/ajcn.2007.25765. Epub 2008 Dec 3. PMID 19056593
- [Result] Kao C, Hsu J, Bandi V, Jahoor F. Alterations in glutamine metabolism and its conversion to citrulline in sepsis. Am J Physiol Endocrinol Metab. 2013 Jun 15;304(12):E1359-64. doi: 10.1152/ajpendo.00628.2012. Epub 2013 Apr 23. PMID 23612995
- [Result] Wijnands KA, Vink H, Briede JJ, van Faassen EE, Lamers WH, Buurman WA, Poeze M. Citrulline a more suitable substrate than arginine to restore NO production and the microcirculation during endotoxemia. PLoS One. 2012;7(5):e37439. doi: 10.1371/journal.pone.0037439. Epub 2012 May 29. PMID 22666356
- [Result] Ware LB, Magarik JA, Wickersham N, Cunningham G, Rice TW, Christman BW, Wheeler AP, Bernard GR, Summar ML. Low plasma citrulline levels are associated with acute respiratory distress syndrome in patients with severe sepsis. Crit Care. 2013 Jan 17;17(1):R10. doi: 10.1186/cc11934. PMID 23327349
- [Result] Cynober L. Citrulline: just a biomarker or a conditionally essential amino acid and a pharmaconutrient in critically ill patients? Crit Care. 2013 Mar 11;17(2):122. doi: 10.1186/cc12534. PMID 23509945